CLINICAL TRIAL: NCT02407210
Title: A Phase 3, Double-Blind, Randomized, Parallel-Group Study to Evaluate the Efficacy and Safety of Azilsartan Compared to Olmesartan Medoxomil in Chinese Participants With Grade I or II Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan Compared to Olmesartan Medoxomil in Chinese Participants With Grade I or II Essential Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-AQST-2014
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-01

CONDITIONS: Essential Hypertension
Keywords: Azilsartan，Olmesartan Medoxomil
MeSH Terms: conditions — Essential Hypertension | interventions — azilsartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- azilsartan group (Experimental): Once-daily oral administration of 20 or 40 mg tablet before or after breakfast
  Interventions: Drug: azilsartan
- olmesartan medoxomil group (Active Comparator): Once-daily oral administration of 20 or 40 mg tablet before or after breakfast
  Interventions: Drug: Olmesartan medoxomil

INTERVENTIONS:
Drug: azilsartan
  Arms: azilsartan group
Drug: Olmesartan medoxomil
  Arms: olmesartan medoxomil group

SUMMARY:
To investigate the efficacy and safety of azilsartan compared to olmesartan medoxomil in patients with grade I or II essential hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes. eighteen years or older and no more than 70 years at the time of informed consent
2. Grade I or II essential hypertension
3. Both sitting systolic and diastolic blood pressures at Week 0 during the run-in period meet the following criteria:

   Sitting systolic blood pressure: greater than or equal to 150 mmHg and less than 180 mmHg

   Sitting diastolic blood pressure: greater than or equal to 95 mmHg and less than 110 mmHg
4. Able to understand the content of the study and comply with the study and to give informed consent in writing before participating in the study

Exclusion Criteria:

1. Secondary hypertension, grade III hypertension (sitting systolic blood pressure greater than or equal to 180 mmHg or sitting diastolic blood pressure greater than or equal to 110 mmHg), or malignant hypertension，hypertensive emergencies，hypertensive urgencies
2. The following circulatory-related diseases or symptoms:

(1) Cardiac disease: angina pectoris; valvular stenosis; atrial fibrillation; the following diseases requiring medication: congestive heart failure or arrhythmia； (2) Cerebrovascular disorder: cerebral infarction, cerebral hemorrhage (onset within 24 weeks before start of the screening period), transient ischemic attack (onset of an attack within 24 weeks before start of the screening period)； (3) Vascular disease: arteriosclerosis obliterans with symptoms of intermittent claudication； (4) Progressive hypertensive retinopathy: hemorrhage, exudation, or papilledema (observed within 24 weeks after start of the screening period)

3. Decrease in sitting diastolic blood pressure by 8 mmHg or more at the end of the run-in period (Week 0) compared to the start of the screening period

4. Day/night reversal, e.g., nightshift worker

5. Unilateral or bilateral renal artery stenosis

6. Clinically apparent hepatic and renal impairment (e.g., with AST and ALT values of 2.5 x upper limit of normal or higher, with serum creatinine value of 1.5 x upper limit of normal or higher during the screening period)

7. Hyperkalemia (with a laboratory value of 5.5 mEq/L or higher during the run-in period)

8. Malignant tumor

9. Compliance with the study drug of less than 80% during the run-in period

10. Poorly-controlled diabetes mellitus (fasting plasma glucose greater than 11mmol/L)，and/or complications (kidney disease, peripheral neuropathy) at Screening.

11. History of hypersensitivity or allergy to olmesartan medoxomil tablets and related drugs (ARB, ACE inhibitors, and renin inhibitors)

12. History of drug abuse (defined as illegal drug use) or alcohol dependency within 2 years before start of the screening period

13. Requirement of the excluded treatment

14. Pregnant or lactating women

15. Participation in another clinical trial or post-marketing clinical trial within 30 days before start of the screening period

16. Dangerous machinery operator such as aerial worker，motor vehicle driver

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Trough sitting diastolic blood pressure (change from end of the run-in period to end of the treatment period) | 16 weeks

SECONDARY OUTCOMES:
Trough sitting systolic blood pressure (change from end of the run-in period to end of the treatment period) | 16 weeks
Trough sitting diastolic and systolic blood pressure (change from end of the run-in period to Week 8 of the treatment period) | 8 weeks
Trough sitting diastolic and systolic blood pressures at each evaluation | 2 weeks
responder rate; rate of patients with normalized blood pressure | 8 weeks and 16 weeks
  Responder is defined as a ≥20mmHg decrease in sitting trough SBP and a ≥10mmHg decrease in sitting trough DBP，or a sitting trough SBP of <140mmHg and a sitting trough DBP of <90mmHg；normalized blood pressure is defined as a sitting trough SBP of <140mmHg and a sitting trough DBP of <90mmHg.
evaluation by ABPM (1: 24-hour mean change in diastolic and systolic blood pressures, 2: Trough/Peak ratio of diastolic and systolic blood pressures)(change from end of the run-in period to Week 14 of the treatment period) | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing ANZHEN Hospital, Beijing, China